CLINICAL TRIAL: NCT03456453
Title: Social Media HIV Prevention Intervention for High Risk Rural Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R34DA045563-01A1 (NIH); 1R34DA045563-01A1 (NIH)
Record Dates: First submitted 2018-02-17; First posted 2018-03-07 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIDA Standard via Facebook (Experimental): Participants will receive the NIDA Standard via Facebook
  Interventions: Behavioral: NIDA Standard for HIV Prevention
- Re-entry services as usual (No Intervention): Participants will receive standard re-entry services available in the community and through the criminal justice system

INTERVENTIONS:
Behavioral: NIDA Standard for HIV Prevention — The NIDA Standard is a manualized, HIV prevention education intervention focused on reducing risky sexual and drug use practices. It will be adapted for Facebook in this pilot trial.
  Arms: NIDA Standard via Facebook

SUMMARY:
The overall aim of this R34 application is to adapt and feasibility test an evidence-based HIV prevention education for high-risk, underserved rural women in Appalachia. This study has potential to make a significant contribution to science by advancing knowledge on the use of social media to increase access to prevention interventions to reduce high-risk substance use and related health disparities among rural women during a time of emerging and significant public health risk in Appalachia. Successfully accomplishing study aims will respond to a critical and unmet need to increase access to prevention interventions using social media, as well as advance knowledge about the high-risk drug use behaviors among vulnerable populations.

DETAILED DESCRIPTION:
The overall aim of this R34 application is to adapt and feasibility test an evidence-based intervention for HIV prevention for a high-risk group of rural women in Appalachia. This study has potential to make a significant contribution to science by advancing knowledge on the use of social media to increase access to prevention interventions to reduce high-risk substance use and related health disparities among rural women during a time of emerging and significant public health risk in Appalachia. Successfully accomplishing study aims will respond to a critical and unmet need to increase the reach and scope of prevention interventions using social media, as well as advance knowledge about the high-risk drug use behaviors of this underserved group. Considering the need for prevention interventions among this high-risk group and the popularity of Facebook, the purpose of this R34 proposal is to adapt an evidence-based HIV prevention intervention for social media delivery and to feasibility test through a randomized control trial with 60 high-risk rural women drug users. The following aims guide the proposed study: (1) Adapt the NIDA Standard for HIV prevention for delivery via Facebook; and (2) Examine the feasibility of the adapted intervention with high-risk rural women through a randomized control pilot. The proposed use of Facebook in this study is promising because it is a stable, widely used, cost-efficient platform that could be leveraged to increase access to critically needed HIV prevention education. This study presents an exciting opportunity to examine the use of Facebook as a technique to expand the reach of evidence-based preventions interventions for high-risk drug users who are not likely to engage in formal treatment. Findings from this study will inform development of the larger R01 which would allow examination of the effectiveness and sustainability of this HIV prevention intervention in understudied, high risk populations.

ELIGIBILITY:
Inclusion Criteria:

* NM-ASSIST indicators of high-risk drug use during the 6 months before jail (including injection);
* engagement in at least one sexual risk behavior in the past 3 months;
* no evidence of cognitive impairment (GAIN, Dennis, 1998),
* no evidence of active psychosis (currently experiencing hallucinations),
* no self-reported current symptoms of physical withdrawal from a recent episode of drug use;
* self-reported HIV negative status;
* projected jail release date within 3 months;
* active Facebook user prior to entering jail (defined as having a Facebook account that was checked at least once a week); and
* reside in a rural, Appalachian county prior to incarceration.

Exclusion Criteria:

* Not incarcerated and screened eligible based on above mentioned criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of being female
Enrollment: 60 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Staton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NIDA Standard Via Facebook | Re-entry Services as Usual
Started | 30 | 30
Completed | 27 | 23
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Not released to community | 1 | 5
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIDA Standard Via Facebook | Re-entry Services as Usual | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Individuals who completed follow-up interviews were included
  years | 34.6 (8.6) | 38.3 (7.3) | 36.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of Years of Education Completed [Mean (Standard Deviation); unit: years] — Population: Individuals who completed follow-up interviews were included
  years | 11.6 (2.0) | 12.7 (1.9) | 12.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Facebook Enrollment
Description: The number of participants who are released and accept the "friend" request from the Facebook study profile
Time Frame: 3 months
Population: Number of participants released from jail, thus eligible to accept the "friend" request from the Facebook profile. All participants who were released were eligible to accept the "friend" request then individuals randomized to the NIDA Standard via Facebook were sent an additional invite to the closed intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | NIDA Standard Via Facebook | Re-entry Services as Usual
Number analyzed (Participants) | 29 | 25
Participants | 15 | 15

2. Secondary Outcome: Number of Participants With Use of Injected Drugs
Description: Use of injected drugs in the last 3-months at follow-up
Time Frame: 3 months
Population: Individuals who were released and completed the 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | NIDA Standard Via Facebook | Re-entry Services as Usual
Number analyzed (Participants) | 27 | 23
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: 3 months after Baseline completion
Description: Adverse event information was only collected at the 3 month follow up
Arm/Group | NIDA Standard Via Facebook | Re-entry Services as Usual
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/23
Other Adverse Events (participants affected / at risk) | 20/27 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIDA Standard Via Facebook (N=27) | Re-entry Services as Usual (N=23)
Non-fatal overdose (General disorders) | 2 | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIDA Standard Via Facebook (N=27) | Re-entry Services as Usual (N=23)
Reincarcerated (Social circumstances) | 8 | 7
Any health problems (General disorders) | 10 | 11
Any mental health problems (Psychiatric disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT03456453/Prot_SAP_ICF_000.pdf